CLINICAL TRIAL: NCT06127381
Title: An Open-label Study of the Safety and Pharmacokinetics of the Glycolic Acid Tetrasubstituted Piceatannol (TGKP, "Study Drug") With a Single Intravenous Administration With Participation of Healthy Volunteers: 3 Arms With Dose Escalation
Brief Title: An Open-label Study of the Safety and Pharmacokinetics of the TGKP
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Gamaleya Research Institute of Epidemiology and Microbiology, Health Ministry of the Russian Federation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 01-TGKP-2023
Record Dates: First submitted 2023-11-07; First posted 2023-11-13 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Acute Respiratory Distress Syndrome (ARDS)
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1/4 therapeutic dose (TGKP) (Experimental): First 5 (five) healthy volunteers will receive (a single intravenous administration) 1/4 therapeutic dose.
  Before administration the study drug will be dosed and diluted in 200 ml of isotonic solution of 0.9% sodium chloride, and then will be administered once intravenously via infusion.
  Interventions: Drug: Glycolic acid tetrasubstituted piceatannol (TGKP)
- 1/2 therapeutic dose (TGKP) (Experimental): Next 5 (five) healthy volunteers will receive (a single intravenous administration) 1/2 therapeutic dose.
  Before administration the study drug will be dosed and diluted in 200 ml of isotonic solution of 0.9% sodium chloride, and then will be administered once intravenously via infusion.
  Interventions: Drug: Glycolic acid tetrasubstituted piceatannol (TGKP)
- Full therapeutic dose (TGKP) (Experimental): Next 15 (fifteen) healthy volunteers will receive (a single intravenous administration) the full therapeutic dose.
  Before administration the study drug will be dosed and diluted in 200 ml of isotonic solution of 0.9% sodium chloride, and then will be administered once intravenously via infusion.
  Interventions: Drug: Glycolic acid tetrasubstituted piceatannol (TGKP)

INTERVENTIONS:
Drug: Glycolic acid tetrasubstituted piceatannol (TGKP) — A total of 25 volunteers will be randomized and receive the study drug, of which 5 - will receive ¼ therapeutic dose, 5 - will receive ½ therapeutic dose, 15 - will receive the full therapeutic dose.

SUMMARY:
The purpose of the trial is to study the tolerability, safety and pharmacokinetics of the study drug with participation of healthy volunteers after single intravenous administration with dose escalation (0.03 mg/kg, 0.06 mg/kg and 0.12 mg/kg).

Before administration the study drug will be dosed and diluted in 200 ml of isotonic solution of 0.9% sodium chloride, and then will be administered once intravenously via infusion.

During the entire follow-up period, the effect of the study drug on vital signs, instrumental and laboratory data, the development, severity and association of adverse events with the study drug will be monitored, investigated and studied.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent to participate in the study;
2. Men and women aged 18 to 45;
3. Healthy volunteers according to the results of a medical examination: no history, as well as according to a screening examination, of pathologies from the gastrointestinal tract, liver, kidneys, cardiovascular system, central nervous system, musculoskeletal system, genitourinary, immune and endocrine systems, blood, which may affect the safety of the volunteer and the assessment of the results of the study (clinical, instrumental and laboratory studies did not reveal diseases or clinically significant abnormalities);
4. Body mass index from 19 to 30;
5. Negative test result for HIV, hepatitis, syphilis;
6. Negative test for the presence of narcotic and psychostimulant drugs in the urine;
7. Negative alcohol test;
8. Negative pregnancy test (for women of childbearing age);
9. Indicators of general and biochemical blood tests at screening within 1.1 x (upper limit of the reference interval) - 0.9 x (lower limit of the reference interval);
10. Consent to the use of barrier contraception methods by the volunteer and his partner during the study period and for 3 months after it.

Exclusion Criteria:

A volunteer may terminate his participation in the study at any stage of its implementation. The principal investigator may remove a volunteer from the study at any time in the following cases:

1. The researcher decided that the volunteer must be excluded in the interests of the volunteer himself.
2. The volunteer is uncooperative or undisciplined.
3. The volunteer was included in violation of the rules of the Protocol.
4. The volunteer needs additional treatment.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Occurrence of AE | Within 28 days after administration of the drug
  Occurrence of adverse events (AE)
Occurrence of SAEs | Within 28 days after administration of the drug
  Occurrence of serious adverse events (SAEs)

IPD SHARING:
Plan to Share IPD: No